CLINICAL TRIAL: NCT04422314
Title: ImmuneSense Lyme Study
Status: Completed | Type: Observational
Sponsor: Adaptive Biotechnologies (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-00717
Record Dates: First submitted 2020-06-01; First posted 2020-06-09 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Lyme Disease
Keywords: erythema migrans rash; bullseye rash; early acute Lyme disease
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Cohort 1: Lyme disease testing cohort
  Interventions: Diagnostic Test: T-Detect Lyme
- Cohort 2: Endemic, asymptomatic controls
  Interventions: Diagnostic Test: T-Detect Lyme
- Cohort 3: Non-endemic, asymptomatic controls
  Interventions: Diagnostic Test: T-Detect Lyme
- Cohort 4: Potential cross-reactive disease states
  Interventions: Diagnostic Test: T-Detect Lyme
- Cohort 5: Lyme disease testing cohort
  Interventions: Diagnostic Test: T-Detect Lyme

INTERVENTIONS:
Diagnostic Test: T-Detect Lyme — T-Detect Lyme is an investigational use test that uses multiplex PCR and NGS to assess rearranged T-cell receptor beta (TRB) gene sequences from genomic DNA isolated from human peripheral blood.

SUMMARY:
ImmuneSense Lyme is a study, which is designed to better understand the immune response to Lyme disease. This is critically important because the immune system may be able to tell us important information about how our own bodies detect and respond to the disease that current tests cannot. Data collected from this study may accelerate the development of better diagnostics for Lyme disease and improve outcomes for many.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* Participants at or above the age of 7
* Arm A: Participants with an EM rash ≥ 5 cm (confirmed by Lyme disease independent expert) with or without other signs and symptoms of Lyme disease
* Arm B: Participants who do not have an EM rash >/= 5 cm (either not confirmed by a Lyme disease independent expert or lacking a rash), but who have signs and symptoms suggestive of Lyme disease that warrants further testing, such as, but not limited to fever, myalgias, malaise, lymphadenopathy, rigors, arthralgias, peripheral and radiculoneuropathy, encephalopathy, intermittent arthritis, meningitis, heart block, carditis, etc

Cohort 2:

- Individuals in general good health, who reside in Lyme disease endemic regions

Cohort 3:

- Individuals in general good health, who reside in a region that is non-endemic for Lyme disease

Cohort 4:

Sourced from a sample repository

* Biorepositories with documented consent from participants for secondary use of their sample by a third party
* Confirmed, documented diagnoses for one of the following diseases:
* Viral: Epstein-Barr virus (EBV), cytomegalovirus (CMV), influenza, or COVID-19
* Tick-borne diseases: babesiosis, rocky mountain spotted fever, anaplasmosis, or ehrlichiosis
* Bacterial infection: syphilis
* Autoimmune/rheumatologic/neurologic diseases: Systemic Lupus Erythematous (SLE), Rheumatoid Arthritis (RA), Multiple Sclerosis (MS), chronic fatigue syndrome
* For infections, active infections are preferred and should be prioritized. Past infections will be acceptable for infections that are difficult to obtain.

Prospective collection Inclusion criteria

* Confirmed, documented diagnoses for one of the following diseases:
* Viral: Epstein-Barr virus (EBV), cytomegalovirus (CMV), influenza, or COVID-19
* Tick-borne diseases: babesiosis, rocky mountain spotted fever, anaplasmosis, or ehrlichiosis
* Bacterial infection: syphilis
* Autoimmune/rheumatologic/neurologic diseases: Systemic Lupus Erythematous (SLE), Rheumatoid Arthritis (RA), Multiple Sclerosis (MS), or chronic fatigue syndrome
* For infections, active infections are preferred and should be prioritized. Past infections will be acceptable for infections that are difficult to obtain.

Cohort 5:

* Participants ages 18 and above
* Arm A: Participants with an EM rash ≥ 5 cm (confirmed by Lyme disease independent expert) with or without other signs and symptoms of Lyme disease
* Arm B: Participants who do not have an EM rash >/= 5 cm (either not confirmed by a Lyme disease independent expert or lacking a rash), but who have signs and symptoms suggestive of Lyme disease that warrants further testing, such as, but not limited to fever, myalgias, malaise, lymphadenopathy, rigors, arthralgias, peripheral and radiculoneuropathy, encephalopathy, intermittent arthritis, meningitis, heart block, carditis, etc

Exclusion Criteria:

* Participants will be excluded from the study if they meet any of the following criteria:
* Participant is a pregnant woman, prisoner, mentally disabled person, or ward-of-the state.
* Participant has any significant condition, laboratory abnormality, or psychiatric illness that would prevent the participant from safely participating in the study.
* Participant has been exposed to an investigational drug (new chemical entity) within 60 days prior to enrollment at the discretion of the investigator.
* Participant has donated more than one pint or 500cc of blood in the past two months or weight-based limits for pediatric populations.
* Received the Lyme disease vaccine
* Chronic infection with HIV, Tuberculosis, Hepatitis C, or Hepatitis B
* Active malignancy

Min Age: 7 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants include male and female participants, of any race and ethnicity, ages 7 and above (inclusive) at the time of enrollment. For Cohort 5 only, participants must be 18 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 893 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
To evaluate sensitivity of T-Detect Lyme Assay relative to STTT and MTTT | Baseline
  Diagnostic sensitivity is defined as the percentage of persons who have a given disorder who are identified by the assay as positive for Lyme disease.
To demonstrate Specificity of T-Detect Lyme Assay relative to STTT and MTTT | Baseline
  Diagnostic specificity is defined as the percentage of persons who do not have a given condition who are identified by the assay as negative for Lyme disease.

CONTACTS AND LOCATIONS:
Overall Officials: Namita Singh, MD, Study Director — Medical Director, Clinical Development
Locations (32):
- United States (32):
  - Adaptive Biotechnologies Investigational Site, Danbury, Connecticut
  - Adaptive Biotechnologies Investigational Site, Macon, Georgia
  - Adaptive Biotechnologies Investigational Site, Savannah, Georgia
  - Adaptive Biotechnologies Investigational Site, Baton Rouge, Louisiana
  - Adaptive Biotechnologies Investigational Site, Lewiston, Maine
  - Adaptive Biotechnologies Investigational Site, Elkridge, Maryland
  - Adaptive Biotechnologies Investigational Site, Rockville, Maryland
  - Adaptive Biotechnologies Investigational Site, Towson, Maryland
  - Adaptive Biotechnologies Investigational Site, Beverly, Massachusetts
  - Adaptive Biotechnologies Investigational Site, Methuen, Massachusetts
  - Adaptive Biotechnologies Investigational Site, Springfield, Massachusetts
  - Adaptive Biotechnologies Investigational Site, Freehold, New Jersey
  - Adaptive Biotechnologies Investigational Site, Binghamton, New York
  - Adaptive Biotechnologies Investigational Site, Endwell, New York
  - Adaptive Biotechnologies Investigational Site, New Windsor, New York
  - Adaptive Biotechnologies Investigational Site, Syracuse, New York
  - Adaptive Biotechnologies Investigational Site, Altoona, Pennsylvania
  - Adaptive Biotechnologies Investigational Site, Hatboro, Pennsylvania
  - Adaptive Biotechnologies Investigational Site, Pittsburgh, Pennsylvania
  - Adaptive Biotechnologies Investigational Site, Scottdale, Pennsylvania
  - Adaptive Biotechnologies Investigational Site, Smithfield, Pennsylvania
  - Adaptive Biotechnologies Investigational Site, Tipton, Pennsylvania
  - Adaptive Biotechnologies Investigational Site, Uniontown, Pennsylvania
  - Adaptive Biotechnologies Investigational Site, Warwick, Rhode Island
  - Adaptive Biotechnologies Investigational Site, Dakota Dunes, South Dakota
  - Adaptive Biotechnologies Investigational Site, Rapid City, South Dakota
  - Adaptive Biotechnologies Investigational Site, Burke, Virginia
  - Adaptive Biotechnologies Investigational Site, Danville, Virginia
  - Adaptive Biotechnologies Investigational Site, Norfolk, Virginia
  - Adaptive Biotechnologies Investigational Site, Kingwood, West Virginia
  - Adaptive Biotechnologies Investigational Site, Morgantown, West Virginia
  - Adaptive Biotechnologies Investigational Site, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No